CLINICAL TRIAL: NCT03053544
Title: Metformin With Neoadjuvant Chemoradiation to Improve Pathologic Responses in Rectal Cancer: An Internal Pilot Study
Brief Title: Metformin With Neoadjuvant Chemoradiation to Improve Pathologic Responses in Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Sunnybrook Research Institute (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 472-2015
Record Dates: First submitted 2016-12-20; First posted 2017-02-15 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Rectal Neoplasm Carcinoma in Situ Adenocarcinoma
Keywords: rectal cancer; adenocarcinoma of the rectum; node positive rectal tumors; metformin; neoadjuvant chemoradiation
MeSH Terms: conditions — Rectal Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): Participants will self-administer 500mg metformin twice daily by mouth: 1) beginning 1 to 2 weeks prior to standard of care CRT, 2) during standard of care CRT and 3) until 30 days after the end of standard of care CRT.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Participants will self-administer 500mg metformin twice daily by mouth: 1) beginning 1-2 weeks prior to standard of care CRT, 2) during standard of care CRT and 3) until 30 days after the end of standard of care CRT.

SUMMARY:
This study is a phase II, single arm, controlled, open label internal pilot.

DETAILED DESCRIPTION:
This internal pilot will be the first prospective study to assess the feasibility and efficacy of adding metformin in non-diabetic rectal patients who undergo standard of care neoadjuvant chemoradiation therapy (CRT). The translational aim of the study will inform on predictive factors (such as p53) and mechanism of action (hypoxia, proliferation). Metformin has been used for decades in patients with type 2 diabetes and has an extremely safe toxicity profile. With current interest in the use of metformin as a cancer therapeutic in non-diabetics, this study is expected to provide proof-of principle data for a larger study.

ELIGIBILITY:
Inclusion Criteria:

1. Plan for care inclusive of:

   i. standard of care neoadjuvant chemoradiation ii. planned total mesorectal excision (TME)
2. Histologically confirmed adenocarcinoma of the rectum
3. At least one of the following:

   i. T3 or T4 lesions ii. T2 lesions ≤ 1 mm to the mesorectal fascia iii. Node positive rectal tumor
4. ECOG performance status of 0 or 1
5. Provide written informed consent
6. Female participants of childbearing potential agree to use adequate methods of contraception from the start of metformin administration until the start of CRT. Contraception will not be required to be continued during or after CRT as this treatment renders participants infertile. Clinically acceptable methods of birth control for this study include intrauterine devices (IUD), birth control pills, hormonal implants, injectable contraceptives, and using barrier methods such as condoms, vaginal diaphragm with spermicide, or sponge.

Exclusion Criteria:

1. Diagnosis of diabetes
2. Current use of metformin
3. Prior pelvic radiation
4. Life expectancy < 6 months.
5. Active infection
6. Creatinine > 1.5X ULN, within 1 month prior to baseline
7. AST, ALT > 2.5X ULN, within 1 month prior to baseline
8. Bilirubin > 1.5 ULN, within 1 month prior to baseline
9. Pregnant or breastfeeding women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12-08; Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) rate | 1 year
  The primary outcome is to evaluate the use of metformin to improve pathological complete response (pCR) rates in non-diabetic participants undergoing standard of care neoadjuvant CRT for rectal cancer.
  The primary outcome will be measured by the pathological complete response rate after completion of the study treatment.

SECONDARY OUTCOMES:
Tumor Proliferation Reduction | 1 year
  The secondary outcome is to determine if metformin reduces tumor proliferation in this study population. The secondary outcome will be determined by examining tumor cell proliferation from longitudinal biopsy specimens.
Tumor Hypoxia | 1 year
  The secondary outcome is to determine if metformin reduces tumor hypoxia in this study population. The secondary outcome will be determined by examining tumor cell hypoxia from longitudinal biopsy specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Wong, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Marianne Koritzinsky, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Results from this internal pilot will be disseminated to participants and stakeholders by means of publication and presentation where appropriate.